CLINICAL TRIAL: NCT06119360
Title: Comparison of the Intubation Success Rate Between Two Techniques Using Lightwand in Patients Undergoing Spine Surgery: Conventional vs. Face-to-face Technique
Brief Title: Comparison of Two Different Lightwand Intubation Techniques in Cervical Immobilized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Hyungseok Seo, Assistant professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KHNMC 2018-10-011-002
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Intubation; Difficult or Failed

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Conventional (Other): Conventional approach using group in lightwand intubation
  Interventions: Procedure: Conventional approach
- Group Face-to-Face (Other): Face-to-face approach using group in lightwand intubation
  Interventions: Procedure: Face-to-face approach

INTERVENTIONS:
Procedure: Face-to-face approach — A front-facing approach and insert the lightwand following the patient's tongue base curvature without scooping movement
  Arms: Group Face-to-Face
Procedure: Conventional approach — Patients were positioned supine and the intubator stood above the patient's head. Opening the mouth and slightly pulling the mandible with one hand, the intubator inserted the lightwand-tracheal tube assembly at midline into the patient's mouth under the ambient light being turned off. To identify the location of the lighted tip, the intubator could move the lightwand back and forth gently, Once the red light of the tip was located at the midline of the patient's neck, the pre-launched tube was inserted smoothly into the patient's airway unless there was no resistance
  Arms: Group Conventional

SUMMARY:
This study compares two different approaches of lightwand intubation techniques in cervical immobilized patients.

DETAILED DESCRIPTION:
This study compares two approaches in lightwand intubation techniques in cervical immobilized patients. One is a conventional approach that involves scooping movement with mandible protraction. The other is a face-to-face approach that inserts lightwand with a front-facing position. This study is conducted as a randomized, prospective, single-blinded design.

ELIGIBILITY:
Inclusion Criteria:

* adults with American Society of Anesthesiologists physical status 1-3
* patients who received scheduled spine surgery under general anesthesia

Exclusion Criteria:

* patients with body mass index <18.5 kg/m2 or >35.0 kg/m2,
* patients who previously had head and neck surgery,
* patients who are at high risk of aspiration,
* patients with pathologic conditions such as tumors, polyps, or inflammation in the airway,
* patients who cannot sit due to severe spine deformity,
* patients who have compromised cardiopulmonary function patients with clinically significant neurovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Initial success rate | during intubation
  Intubation success rate at the first attempt

SECONDARY OUTCOMES:
Intubation time | during intubation
  Total time to the successful intubation

OTHER OUTCOMES:
Immediate intubation related outcomes | Immediately after general anesthesia (at the post anesthesia care unit)
  Outcomes after tracheal intubation
24 hours intubation related outcomes | 24 hours after general anesthesia (at the general ward)
  Outcomes after tracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Hyungseok Suh, Principal Investigator — Kyung Hee University Hospital at Gangdong-gu
Locations (1):
- Kyung Hee University Gangdong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No